CLINICAL TRIAL: NCT04858646
Title: Effects of Aerobic Exercises on Gross Motor Function in Children With Spastic Cerebral Palsy
Brief Title: Aerobic Exercises and Gross Motor Function in Spastic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/19/2021 Hira Nawaz
Record Dates: First submitted 2021-03-30; First posted 2021-04-26 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Spastic Cerebral Palsy
Keywords: Cerebral palsy; Gross motor function measure; Aerobic exercises
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic exercises (Experimental): Subjects in A group was treated with different types of aerobic exercises such as 10 minute walking, 10 minute trampoline exercise and 10 minutes ball throwing activities
  Interventions: Other: Experimental( Group A ): Aerobic exercises
- Conventional physical therapy (Active Comparator): Traditional physical therapy The group B was treated with conventional therapy. Conventional treatment protocol passive ROM and stretching passive ROM for 15 minutes and stretching for 15 minutes. Treatment duration for both groups will be 30 minutes. Each subject received total 30 sessions of the treatment, with 5 treatment sessions per week for 6 weeks. Post treatment reading were collected after end of 6th weeks.
  Interventions: Other: Conventional( Group B): Conventional Physical therapy

INTERVENTIONS:
Other: Experimental( Group A ): Aerobic exercises — Subjects in A group was treated with different types of aerobic exercises such as 10 minute walking, 10 minute trampoline exercise and 10 minutes ball throwing activities
  Arms: Aerobic exercises
Other: Conventional( Group B): Conventional Physical therapy — The group B was treated with conventional therapy. Conventional treatment protocol passive ROM and stretching passive ROM for 15 minutes and stretching for 15 minutes.Treatment duration for both groups will be 30 minutes. Each subject received total30sessions of the treatment, with 5 treatment sessions per week for 6 weeks
  Arms: Conventional physical therapy

SUMMARY:
The aim of this research is to find the effects of aerobic exercise on gross motor function in cerebral palsy patients. Quasai experimental study done at Noor Zainab Rehabilitation center, Lahore. The sample size was 34. The subjects were divided in two groups, 17 subjects with aerobic exercise 17 children with conventional treatment. Sampling technique applied was purposive non probability sampling. Only 7-12 years individuals with GMFCS level I- III were included. Tools used in the study were Gross motor function measure (GMFM-66 and 88) .Data was be analyzed through SPSS 21.

DETAILED DESCRIPTION:
Cerebral palsy" an umbrella term for a group of irreversible and non-progressive abnormalities of the fetal or neonatal brain, this can lead to disorders of movement and posture. National Institute for Health and Care Excellence (NICE) states that, it is the most common cause of physical disability in children and young people in the developing world. CP is condition with multiple causes; multiple clinical types; multiple associated developmental pathologies, such as intellectual disability, autism, epilepsy, and visual impairment; and more recently multiple rare pathogenic genetic variations Motor disability in cerebral palsy is related with sitting, standing, walking and running appears as the main symptom in children with CP, the assessment and management of CP have focused on gross motor function. The Gross Motor Function Measure (GMFM) is designed by Russell et al. in 1993 is used to measure the level of motor development and changes of gross motor function in a standardized environment in children with CP. GMFM-66 is comprised of a subset of the 88 items identified as contributing to the measure of gross motor function in children with CP, ranging from 0 (lowest motor function) to 100 (highest motor function). Cardiorespiratory endurance is an integral component of physical fitness and has been identified as the most important fitness component associated with health and mortality. In clinical practice, rebound is usually offered as a 20 minute session, once per week for 6 weeks. Typical rebound therapy programs target gross motor skill development, such as balance while sitting, kneeling, standing and walking; functional transfers such as rolling and sit to stand; aerobic activity such as jumping. It is theorized that using a trampoline improves muscle tone, posture, balance, kinesthetic awareness, movement, body awareness, and communication. Aerobic exercise may improve activity as indicated by motor function but does not appear to improve gait speed, walking endurance, participation or aerobic fitness among children with CP in the short or intermediate term. Researcher to conduct a study on effects of robot assisted gait training in CP children, collect data from 14 consecutive children affected by CP, each session of 60 minutes, 20 daily sessions for 5 days per week. Saeid Fatorehchy et al. in 2019 conducted an RCT, this study was to evaluate the effects of aquatic therapy in cerebral palsy patients. Six children with average age of 7 years 4 months are included. Each sessions lasted for 50 minutes, comprising 10 minutes of warm up and stretching and 40 minutes of walking in pool at different at different water depths.

Maria A. Fragala-Pinkham et al. stated that participation in routine physical activity is important for health promotion and prevention of chronic health condition. Participating in sports and active recreation can be beneficial on several levels for children and adults with CP. At the body function and structure level of the ICF, improvement in fitness and endurance have been documented for children and young with CP. Sports equipment that can be use are cycling, swimming, sketching and outdoor active recreation.

ELIGIBILITY:
Inclusion Criteria:

* Children with CP at GMFCS level I- III

Exclusion Criteria:

* Botulinum toxin-A- injection in lower limb last 6 months
* <0° dorsiflexion in ankle
* Unable to cooperate and follow instructions
* Children with progressive brain disorder

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Gross motor function measure (GMFM-66 and 88) | 3 months
  The Gross Motor Function Measure (GMFM) is an observational clinical tool designed to evaluate change in gross motor function in children with cerebral palsy. There are two versions of the GMFM - the original 88-item measure (GMFM-88) and the more recent 66-item GMFM (GMFM-66) The scoring system of the GMFM is a four-point scale divided into five categories (lying and rolling; sitting; crawling and kneeling; standing; walking, running).

CONTACTS AND LOCATIONS:
Overall Officials: Tehreem Mukhtar, MS, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kwon TG, Yi SH, Kim TW, Chang HJ, Kwon JY. Relationship between gross motor function and daily functional skill in children with cerebral palsy. Ann Rehabil Med. 2013 Feb;37(1):41-9. doi: 10.5535/arm.2013.37.1.41. Epub 2013 Feb 28. PMID 23525125
- [Background] MacLennan AH, Thompson SC, Gecz J. Cerebral palsy: causes, pathways, and the role of genetic variants. Am J Obstet Gynecol. 2015 Dec;213(6):779-88. doi: 10.1016/j.ajog.2015.05.034. Epub 2015 May 21. PMID 26003063
- [Background] Lauglo R, Vik T, Lamvik T, Stensvold D, Finbraten AK, Moholdt T. High-intensity interval training to improve fitness in children with cerebral palsy. BMJ Open Sport Exerc Med. 2016 May 9;2(1):e000111. doi: 10.1136/bmjsem-2016-000111. eCollection 2016. PMID 27900177
- [Background] Kim OY, Shin YK, Yoon YK, Ko EJ, Cho SR. The effect of treadmill exercise on gait efficiency during overground walking in adults with cerebral palsy. Ann Rehabil Med. 2015 Feb;39(1):25-31. doi: 10.5535/arm.2015.39.1.25. Epub 2015 Feb 28. PMID 25750868
- [Background] Balemans AC, Van Wely L, De Heer SJ, Van den Brink J, De Koning JJ, Becher JG, Dallmeijer AJ. Maximal aerobic and anaerobic exercise responses in children with cerebral palsy. Med Sci Sports Exerc. 2013 Mar;45(3):561-8. doi: 10.1249/MSS.0b013e3182732b2f. PMID 23034639
- [Background] Verschuren O, Darrah J, Novak I, Ketelaar M, Wiart L. Health-enhancing physical activity in children with cerebral palsy: more of the same is not enough. Phys Ther. 2014 Feb;94(2):297-305. doi: 10.2522/ptj.20130214. Epub 2013 Oct 3. PMID 24092902
- [Background] Ryan JM, Cassidy EE, Noorduyn SG, O'Connell NE. Exercise interventions for cerebral palsy. Cochrane Database Syst Rev. 2017 Jun 11;6(6):CD011660. doi: 10.1002/14651858.CD011660.pub2. PMID 28602046
- [Background] Digiacomo F, Tamburin S, Tebaldi S, Pezzani M, Tagliafierro M, Casale R, Bartolo M. Improvement of motor performance in children with cerebral palsy treated with exoskeleton robotic training: A retrospective explorative analysis. Restor Neurol Neurosci. 2019;37(3):239-244. doi: 10.3233/RNN-180897. PMID 31177250
- [Background] Gillett JG, Lichtwark GA, Boyd RN, Barber LA. Functional Anaerobic and Strength Training in Young Adults with Cerebral Palsy. Med Sci Sports Exerc. 2018 Aug;50(8):1549-1557. doi: 10.1249/MSS.0000000000001614. PMID 29557839